CLINICAL TRIAL: NCT03176667
Title: Ultrasound Guided Erector Spinae Plane Block in Patients Undergoing Video-assisted Thoracoscopic Surgery (VATS) Lobectomy or Wedge Resections - a Pilot Randomized Control Trial
Brief Title: Ultrasound Guided Erector Spinae Plane Block in Patients Undergoing VATS Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3012
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Post-operative Pain
Keywords: regional, erector spinae block, lobectomy, video-assisted
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP for VATS (Experimental): Erector Spinae plane (ESP) block
  Interventions: Procedure: Ultrasound guided erector spinae plane block
- ICB for VATS (Active Comparator): Intercostal block (ICB)
  Interventions: Procedure: Intercostal block

INTERVENTIONS:
Procedure: Ultrasound guided erector spinae plane block — A high-frequency linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to the T5 spinous process. The trapezius, rhomboid major, and erector spinae muscles will then be identified superficial to the tip of the T5 transverse process. The patient's skin will be anesthetized with 2% lidocaine. A 17-gauge 8-cm needle will be inserted using an in-plane superior-to-inferior approach to place the tip into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process. A total of 30 mL of 0.5% ropivacaine with 5mcg/mL of epinephrine will be injected in 5-mL aliquots through the needle (maximum of 3mg/kg), followed by insertion of a 19-gauge catheter under direct vision 5 cm beyond the needle tip. The catheter will then be secured in place.
  Arms: ESP for VATS
Procedure: Intercostal block — The surgeons will identify the desired rib, and advance the needle at an approximately 20-degree angle until contact with rib is made, the needle is then walked of the inferior border of the rib and advanced slightly to plaice the tip of the needle in the neurovascular bundle. The intercostal nerve blocks will be performed at T4-T11 using 0.25% Marcaine with epinephrine and a volume of 5 ml per block (maximum of 2.5mg/kg) after negative aspiration has been confirmed.
  Arms: ICB for VATS

SUMMARY:
This study will compare ESP block plus patient-controlled analgesia (PCA) to intercostal nerve block plus PCA as post-operative pain control for patients having video-assisted thorascopic surgeries.

DETAILED DESCRIPTION:
Video assisted thoracoscopic surgery (VATS) has become an increasingly popular technique in thoracic surgery with improvement in technology. It provides significant advantages over open thoracotomy procedures including reduced acute pain, reduced mortality, improved post-operative pulmonary function, and shorter hospitalization stays. Nevertheless, there is still considerable amount of post-operative acute pain with VATS lobectomies. Controlling post-operative pain is crucial because increased acute pain has been associated with the development of chronic pain.

Many patients receive either thoracic epidural (TEA) or paravertebral blocks (PVB) to treat post-operative pain in thoracotomy procedures as these techniques remain the gold standard. In contrast to thoracotomy procedures, it is unclear which is the best approach to analgesia is in VATS. A few studies have found no benefit in pain scores, patient satisfaction, pulmonary function, and incidence of side effects when comparing TEA with opioid patient controlled analgesia in VATS. Other studies have found minimal benefit in pain scores with TEA. The PVB has been used as alternative to TEA. One prospective observational study using PVB and continuous intercostal catheter demonstrated lower pain scores in VATS lobectomy. A randomized control trial (RCT) comparing PVB with wound infiltration in VATS lobectomy showed lower pain scores, lower morphine consumption, and higher patient satisfaction. However, both TEA and PVB have potential serious side-effects and complications. Complications of TEA include severe hypotension, epidural abscess, epidural hematomas and spinal cord injury. PVB have less incidence of hypotension but may involve risks like pneumothorax, pleural and vascular puncture, and higher systemic absorption of local anesthetics. PVB is also technically challenging and its spread is not reliable likely due to the presence of the endothoracic fasica. In addition, placement of both TEA and PVB require appropriate discontinuation of anticoagulants. Intercostal nerve blocks have been used as an analgesic alternative to TEA and PVB. One RCT found patients who had received intercostal blocks undergoing bilateral VATS for hyperhidrosis had lower pain scores in the post-anesthesia recovery unit (PACU). A combined retrospective and prospective study examined the analgesic effect and duration of intercostal blocks in patients undergoing VATS. The authors found that intercostal blocks decreased morphine consumption in the first 24 hours and the analgesic effect of the block lasted approximately 16 hours. Intercostal blocks appear to have some analgesic effect in the immediate post-operative period but are short-lived unless a catheter is placed. The standard practice for post-operative pain management for VATS lobectomy at St. Joseph's hospital consists of intercostal blocks performed by the thoracic surgeons at the end of surgery in combination with patient-controlled analgesia (PCA).

A novel regional technique called the Erector Spinae Plane (ESP) block has been recently described. This interfascial block involves ultrasound guided injection of local anesthetics posterior to the erector spinae muscle and superficial to transverse process of thoracic vertebrae at appropriate level. The ESP block appears to target the dorsal and ventral rami of the spinal nerves as they leave the intervertebral foramen. Cadaveric examination of ESP block showed extensive cranial-caudal spread of the block, approximately four dermatomes above and below the site of injection. The ESP block has been successfully applied in multiple clinical settings. For example, several patients suffering from chronic thoracic neuropathic pain achieved significant analgesia after receiving ESP blocks. ESP blocks have also been used as a rescue analgesia for a patient who failed a TEA after thoracotomy. Other applications include ventral hernia repair in abdominal surgery. The simplicity and safety of the ESP block has been proposed as its main advantages. Because it is a superficial interfascial plane block, it is distant from both the spinal cord and pleura. The ESP block is technically an easy to perform under ultrasound guidance due to its superficial location. There is also theoretically less possibility of needle related complications as the transverse process acts as a backstop for needle advancement. A catheter can be placed easily during the ESP block allowing continuous infusion and prolonged analgesia.

Given the importance of providing adequate analgesia in VATS lobectomy and wedge resections and lack of consensus amongst surgeons and anesthesiologists for the optimal analgesic technique, the investigators are proposing a prospective observational study to examine the analgesic efficacy of the ESP block in VATS lobectomy or wedge resections as a potential alternative to TEA, PVB and intercostal blocks. The investigators are hoping the results of this study will provide framework for future larger comparative studies.

ELIGIBILITY:
Inclusion Criteria:

* Elective video-assisted thoracoscopic surgeries (VATS) lobectomies
* Elective video-assisted thoracoscopic surgeries (VATS) wedge resections

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia
* Known allergy to local anesthetics
* Bleeding diathesis
* Use of any anti-coagulants
* Inability to provide informed consent
* Severe kidney or liver disease
* Inability to operate PCA system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Feasibility comparing two regional techniques in VATS surgery which is defined as the number of patients recruited per week. | One week
  Number of patients recruited per week
Number of adverse events (AEs) which can be attributed to the ESP block which is defines as the number of AEs occuring per week. | One week
  Number of adverse events

SECONDARY OUTCOMES:
Pain scores at rest and on movement | Two days post-operatively
  Pain scores will be recorded at intervals
Dermatome distribution to test loss of sensation to pinpricks | Two days post-operatively
  The dermatome distribution on the patient's anterior chest, mid-axillary line and back will be collected using a blunt needle to test for loss of sensation to pinpricks.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi GP, Bonnet F, Shah R, Wilkinson RC, Camu F, Fischer B, Neugebauer EA, Rawal N, Schug SA, Simanski C, Kehlet H. A systematic review of randomized trials evaluating regional techniques for postthoracotomy analgesia. Anesth Analg. 2008 Sep;107(3):1026-40. doi: 10.1213/01.ane.0000333274.63501.ff. PMID 18713924
- [Background] Demmy TL, Curtis JJ. Minimally invasive lobectomy directed toward frail and high-risk patients: a case-control study. Ann Thorac Surg. 1999 Jul;68(1):194-200. doi: 10.1016/s0003-4975(99)00467-1. PMID 10421140
- [Background] Kim JA, Kim TH, Yang M, Gwak MS, Kim GS, Kim MJ, Cho HS, Sim WS. Is intravenous patient controlled analgesia enough for pain control in patients who underwent thoracoscopy? J Korean Med Sci. 2009 Oct;24(5):930-5. doi: 10.3346/jkms.2009.24.5.930. Epub 2009 Sep 23. PMID 19794994
- [Background] Wildgaard K, Petersen RH, Hansen HJ, Moller-Sorensen H, Ringsted TK, Kehlet H. Multimodal analgesic treatment in video-assisted thoracic surgery lobectomy using an intraoperative intercostal catheter. Eur J Cardiothorac Surg. 2012 May;41(5):1072-7. doi: 10.1093/ejcts/ezr151. Epub 2011 Dec 21. PMID 22219442
- [Derived] Horth D, Sanh W, Moisiuk P, O'Hare T, Shargall Y, Finley C, Hanna W, Agzarian J, Forero M, Davis K, Vanniyasingam T, Thabane L, Shanthanna H. Continuous erector spinae plane block versus intercostal nerve block in patients undergoing video-assisted thoracoscopic surgery: a pilot randomized controlled trial. Pilot Feasibility Stud. 2021 Feb 24;7(1):56. doi: 10.1186/s40814-021-00801-7. PMID 33627193